CLINICAL TRIAL: NCT01079416
Title: Is Capsule Endoscopy Accurate and Cost-effective Enough to Screen Cirrhotic Patients for Varices & Other Lesions?
Brief Title: Study of Capsule Endoscopy to Determine the Accuracy for Detection of Esophageal Varices
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Disaya Chavalitdhamrong, MD, University of California, Los Angeles
Other Study IDs: 01-11-047-12; K24DK002650 (NIH)
Record Dates: First submitted 2010-03-01; First posted 2010-03-03 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: Esophageal Varices
Keywords: Esophageal Capsule Endoscopy, Screening
MeSH Terms: conditions — Esophageal and Gastric Varices | interventions — Endoscopy; Endoscopy, Digestive System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Capsule endoscopy: Study device
  Interventions: Device: Capsule endoscopy, Esophagogastroduodenoscopy
- Esophagogastroduodenoscopy: Gold standard
  Interventions: Device: Capsule endoscopy, Esophagogastroduodenoscopy

INTERVENTIONS:
Device: Capsule endoscopy, Esophagogastroduodenoscopy

SUMMARY:
Esophageal capsule endoscopy is sedation-less alternative to upper endoscopy for evaluating esophageal lesions and potentially other upper gastrointestinal lesions. The purpose of this study was to determine whether esophageal capsule endoscopy is convenient and accurate as upper endoscopy for detection of esophageal varices and related lesions.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years and less than 86 years at the time of consent.
* Clinically evident or biopsy proven cirrhosis.
* No previous documented UGI bleeding due to peptic ulcers, varices, portal hypertensive gastropathy, angiomas, or watermelon stomach.
* No previous endoscopic, radiological or surgical treatment for variceal bleeding or ascites.
* Probable life expectancy of at least 24 months without liver transplantation, as judged by the hepatologist and endoscopist-investigators, and have a Model for End-Stage Liver Disease (MELD) score ≤ 29.
* Signed a written informed consent.

Exclusion Criteria:

* Prior variceal bleeding- esophageal, gastric, or other site.
* Prior endoscopic (e.g. sclerotherapy, ligation, or combination therapy), radiological (e.g. transjugular intrahepatic portosystemic shunt-TIPS) or surgical (e.g. portocaval or splenorenal shunt) treatment of esophagogastric varices or ascites.
* Patient who was uncooperative or unable to give written consent.
* Severe co-morbid illness, e.g. end stage chronic renal disease (e.g. dialysis dependence, creatinine greater than 2 times normal) or respiratory failure (e.g. ventilator dependent, oxygen dependent, unstable asthma or chronic obstructive pulmonary disease- e.g. 2 or more hospitalizations for exacerbation in 1 year, asthma or obstructive pulmonary disease which required daily bronchodilators and/or oral/inhaled steroids), tense ascites requiring repeated therapeutic paracenteses, severe hepatic encephalopathy, peritonitis, or sepsis.
* Active cancer with less than a 24 month expected survival and/or cancer on active treatment with chemotherapy and/or radiation therapy.
* Esophageal motility disorder, esophageal stricture or esophageal diverticulum, causing dysphagia or requiring dilatation.
* GI obstruction or partial obstruction (by history or imaging), symptomatic GI stricture or pseudo-obstruction which may prevent passage of the capsule.
* Patients with potentially reversible portal hypertension such as alcoholic hepatitis, acute viral hepatitis, untreated autoimmune hepatitis, or chronic hepatitis B or C on viral therapy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cirrhotic patients
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2006-06; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
The accuracy of capsule endoscopy for detecting esophageal varices | June 2006-February 2008

SECONDARY OUTCOMES:
Time to perform and interpret capsule endoscopy study | June 2006-February 2008

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA, Los Angeles, California, United States

REFERENCES:
- [Background] Jensen DM. Endoscopic screening for varices in cirrhosis: findings, implications, and outcomes. Gastroenterology. 2002 May;122(6):1620-30. doi: 10.1053/gast.2002.33419. PMID 12016427
- [Background] Jutabha R, Jensen DM, Martin P, Savides T, Han SH, Gornbein J. Randomized study comparing banding and propranolol to prevent initial variceal hemorrhage in cirrhotics with high-risk esophageal varices. Gastroenterology. 2005 Apr;128(4):870-81. doi: 10.1053/j.gastro.2005.01.047. PMID 15825071